CLINICAL TRIAL: NCT06828406
Title: Improving Safety, Patient Experience, and Equity Through Shared Decision-making Huddles in Labor (I'M SPEAKING)
Brief Title: Improving Safety, Patient Experience and Equity Through Shared Decision-making Huddles in Labor
Acronym: I'M SPEAKING
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Endeavor Health (Other)
Collaborators: University of Illinois at Chicago (Other); University of Chicago (Other); Ariadne Labs (Other); University of Michigan (Other); Northwestern University (Other); Patient-Centered Outcomes Research Institute (Other)
Responsible Party: Principal Investigator, Ann Borders, Co-Principal Investigator, Endeavor Health
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: Study00000033; BPS-2023C2-33453 (Other Grant/Funding Number: Patient Centered Outcomes Research Institute (PCORI))
Record Dates: First submitted 2024-12-05; First posted 2025-02-14 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-02

CONDITIONS: Perinatal Decision Making
Keywords: Shared Decision Making; Quality Improvement; Cesarean Birth; Labor and Delivery; Nulliparous Term Singleton Vertex; Illinois Perinatal Quality Collaborative; Promoting Vaginal Birth; Birth Equity; Severe Maternal Morbidity

STUDY DESIGN:
Intervention Model Description: Complete Randomized Stepped Wedge Design
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention TeamBirth (Other): shared decision making in labor using team huddles
  Interventions: Behavioral: TeamBirth
- Usual Care (No Intervention): Usual Care

INTERVENTIONS:
Behavioral: TeamBirth — TeamBirth
  Arms: Intervention TeamBirth

SUMMARY:
To evaluate the effectiveness of an existing quality improvement (QI) training program known as TeamBirth, using a randomized stepped-wedge hybrid type II study design, to (a) decrease nulliparous term singleton vertex (NTSV) cesarean birth (CB) across all birthing people, and specifically for Black birthing people, and (b) increase shared decision-making (SDM), (c) improve patient experience of respectful care. TeamBirth uses a train-the-trainer model to implement patient-participatory shared decision-making on Labor and Delivery (L&D) units, with the goal of decreasing unwanted and unnecessary interventions and improving patient experiences and outcomes for labor and birth.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 or older
* English or Spanish speaking
* Gave birth to a live-born infant after laboring

Exclusion Criteria:

* Speaks a language other than English or Spanish
* Under the age of 18
* Gave birth to a nonliving infant
* Cesarean delivery without labor

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 2200 (Estimated)
Dates: Start 2025-04-29 (Actual); Primary Completion 2027-10-31 (Estimated); Study Completion 2029-07 (Estimated)

PRIMARY OUTCOMES:
Nulliparous Term Singleton Vertex (NTSV) Cesarean Birth (CB) | 6 months prior to TeamBirth, 3 months post TeamBirth implementation
  NTSV CB Rate for all birthing people in participating hospitals
Shared Decision Making (SDM) | 6 months prior to TeamBirth, 3 months post TeamBirth implementation
  Childbirth Options, Information, and Person-Centered Explanation (CHOICEs) scale, scores range from 14 to 90, high scores indicate higher levels of shared decision making

SECONDARY OUTCOMES:
NTSV CB in Black birthing people | 6 months prior to TeamBirth , 3 months post TeamBirth implementation
  NTSV CB Rate Black birthing people in participating hospitals
SDM in Black birthing people | 6 months prior to TeamBirth, 3 months post TeamBirth implementation
  Childbirth Options, Information, and Person-Centered Explanation (CHOICEs) scale, scores range from 14 to 90, high scores indicate higher levels of shared decision making
Patient Experience | 6 months prior to TeamBirth, 3 months post TeamBirth implementation
  Illinois Perinatal Quality Collaborative (ILPQC) Patient-Reported Experience Measure (PREM), there is no numerical value assigned to the ILPQC PREM
Patient Experience | 6 months prior to TeamBirth, 3 months post TeamBirth implementation
  Mother's Autonomy in Decision Making (MADM), scores range from 7 to 42, higher scores indicate the women had greater agency and autonomy when engaging in a shared decision making process with a maternity care provider
Patient Experience | 6 months prior to TeamBirth, 3 months post TeamBirth implementation
  Person-Centered Maternity Care Scale for use in the United States (PCMC-US), scores range from 0 to 100, higher scores indicate more person-centered maternity care
Patient Experience | 6 months prior to TeamBirth, 3 months post TeamBirth implementation
  CollaboRATE, scores range from 0 to 100, a higher score means the number of core dimensions of shared decision making are met
Patient Experience | 6 months prior to TeamBirth, 3 months post TeamBirth implementation
  Acceptability of Intervention Measure (AIM), scores range from 3 to 15, the lower the score, the more satisfied the patient was with their care

CONTACTS AND LOCATIONS:
Overall Officials: Ann Borders, Principal Investigator — Endeavor Health; Beth Plunkett, Principal Investigator — Endeavor Health
Locations (1):
- Endeavor Health Evanston Hospital, Evanston, Illinois, United States

IPD SHARING:
Plan to Share IPD: Yes
Data to be banked may include:
  * De-identified transcripts of clinician, birthing person, partner/support person focus groups or interviews
  * De-identified ethnographic field notes
  * De-identified birthing person, partner/support person survey data
  * De-identified administrative data on birth outcomes for Illinois hospitals
Supporting Information: Study Protocol, CSR
Time Frame: 7 years post completion of the final research report. We anticipate the final research report to be completed 7/1/2030.
Access Criteria: Data collected from this study will be de-identified and banked for further use as required by the funder's Policy for Data Management and Data Sharing policy accessible here: https://www.pcori.org/about/governance/pcoris-policy-data-management-and-data-sharing. According to the funder's policy, the full de-identified, cleaned dataset must be maintained for at least 7 years following completion of the final research report to the funder.
URL: https://www.pcori.org/about/governance/pcoris-policy-data-management-and-data-sharing